CLINICAL TRIAL: NCT05498064
Title: A Real World Study of Ensartinib in Advanced ALK-positive Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Real World Study of Ensartinib in Advanced ALK-positive NSCLC
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Wang mengzhao, Chief Director of Department of Respiratory and Critical Care Medicine, Peking Union Medical College Hospital
Other Study IDs: BD-EN-IV007
Record Dates: First submitted 2022-05-17; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Anaplastic Lymphoma Kinase I1171N; Ensartinib
Keywords: Carcinoma, Non-Small-Cell Lung; Anaplastic Lymphoma Kinase; Ensartinib; Real world study
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ensartinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ensartinib — Ensartinib 225 mg administered once daily orally

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of Ensartinib in advanced ALK-positive non-small cell lung cancer, and the mechanisms of population pharmacokinetics and resistance to Ensartinib.

DETAILED DESCRIPTION:
Participants will receive Ensartinib at 225 mg orally once a day (QD). Treatments will continue until disease progression, meeting one of treatment discontinuation criteria (eg, patient decision, adverse event, pregnancy). At the time of disease progression, participants will enter a survival follow-up until death, withdrawal of consent or study closure, whichever occurs earlier. Collection of venous blood sample from participants included 3 times: before treatment, 8 weeks of treatment, and disease progression. Blood specimens of 8 ml were collected each time for ctDNA NGS testing, and evaluation of Ensartinib population pharmacokinetics with blood sampling after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed stage III b or IV NSCLC, according to the International Association for the Study of Lung Cancer staging manual in Thoracic Oncology, 8th edition.
2. Documented ALK-positive disease according to FISH , Ventana IHC ,RT-PCR or NGS;
3. Patients must have demonstrated progression during or after ALK-TKI treatment;
4. Eastern cooperative oncology group performance status (ECOG PS) of 0-2, overall survival>3 months;
5. Patients need radiotherapy or can receive radiotherapy, such as bone metastatic lesions, intrapulmonary lesions, adrenal lesions, etc.
6. Initially general blood tests including complete blood count, biochemistry, electrolytes, and urine biochemistry were performed as a routine screening in order to identify any abnormalities.
7. Male and female patients must agree to abstain or to use two highly effective forms of contraception during the treatment period and for 90 days after the last dose of study medication.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically or cytologically confirmed stage III b or IV NSCLC with ALK -rearrangement
Sampling Method: Non-Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 36 months
  Defined as time from first dose of Ensartinib to disease progression or death due to any causes

SECONDARY OUTCOMES:
The objective response rate (ORR) | 36 months
  ORR per RECIST 1.1 calculated as the proportion of patients with a best overall response defined as complete response (CR) or partial response (PR).
Overall survival (OS) | 48 months
  OS, defined as time from first dose of Ensartinib to death due to any cause
12 month/24 month/36 month/48 month-overall survival (OS) rate OS | 12 months，24 months，36 months，48 months
  Defined as the time from randomization to death from any cause. The OS rate was estimated based on the landmark analysis.
Incidence of patients experiencing adverse events (AE) | 36 months
  Adverse events are graded according to CTCAE 5.0

OTHER OUTCOMES:
Peak plasma concentration (Cmax) of Ensartinib. | Three hours after Ensartinib treatment
  Evaluation of Ensartinib population Cmax pharmacokinetics.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory and Critical Care Medicine, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No